CLINICAL TRIAL: NCT00482157
Title: Calcitriol or Placebo in Men for Prostate Cancer Active Surveillance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROS0022; 97408 (Other: SU IRB)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin D; Calcitriol

INTERVENTIONS:
Drug: Vitamin D (Calcitriol)

SUMMARY:
After the diagnosis of prostate cancer, many men alter their lifestyle or diet or use various supplements in an attempt to retard the growth of their cancer. While there is limited data on the use of diet and supplements to alter the risk of prostate cancer, even less is known regarding the ability of diet or supplements to alter progression. For men who have elected active surveillance, the investigators propose to investigate the ability of vitamin D to retard the growth of prostate cancer.

DETAILED DESCRIPTION:
Men will be randomized to each of two arms for a total of 24 subjects: calcitriol alone (DN101, 45 micrograms once weekly) or placebo. Baseline laboratory assays, including serum PSA, serum and urine calcium and creatinine, will be performed and the EPIC questionnaire (expanded prostate cancer index composite, validated HRQOL tool for prostate cancer patients) will be completed. Patients will also undergo prostate needle biopsy [4 cores taken under transrectal ultrasound (TRUS) guidance] to establish baseline levels of gene expression. Follow-up at the end of 2 weeks (just prior to the third dose) will include a history and physical, and a repeat of all baseline blood and urine tests. Follow-up at 3 months will include a history and physical, repeating all blood and urine tests, and the EPIC questionnaire. At 6 months, in addition to the history and physical, blood and urine tests, and the EPIC questionnaire, a TRUS-guided prostate needle biopsy will be performed. This will be a standard 12-core scheme and 4 of these cores will be used for laboratory analysis. Renal ultrasounds will again be performed on men in the calcitriol arms to look for stones. Patients who show no evidence of clinical progression will be offered to remain on study, in their designated treatment arm, for an additional 6 months. Any patient exhibiting clinical progression at any time will be withdrawn from the study and offered standard treatment options. For patients remaining on study at 12 months, an end-of-study biopsy will be requested (12-core scheme with 4 cores used for laboratory analysis)

ELIGIBILITY:
Inclusion Criteria:- Untreated prostate adenocarcinoma by an extended biopsy (>8 needle cores on systematic prostate biopsy) within 1 year of the screening date

* PSA <10.0 ng/ml
* Gleason sum 6 or <2 mm Gleason pattern 4
* No more than 33% of biopsy cores positive Exclusion Criteria:- Prior or concurrent treatment for prostate cancer
* Use of Finasteride, Dutasteride, Saw Palmetto
* Use of NSAIDs, COX-2 inhibitors and/or aspirin, soy or vitamin D supplements for more than 7 days over the one month prior to study
* Kidney disease, hypercalcemia or renal stones
* ECOG performance status >1
* Uncontrolled hypertension, unstable angina, history of transient ischemic attack (TIA), history of stroke.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
changes in expression of biomarkers as assessed by prostate biopsy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Presti Jr., Principal Investigator — Stanford University